CLINICAL TRIAL: NCT00701298
Title: Inhibition of DNA Methylation by 1-Hr Infusion of 5-aza-2'-Deoxycitidine (Decitabine) x 10 Days (M-F) With Escalating Doses of Sub-Q Pegylated (PEG) Interferon-alpha 2B (PEG-Intron): A Phase I Study With Molecular Correlates
Brief Title: Decitabine With or Without Interferon Alfa-2b in Treating Patients With Unresectable or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00295; NCI-2009-00295 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000597624; NVCI-0725; NVCI 07-25 (Other: Nevada Cancer Institute-Summerlin Campus); 8224 (Other: CTEP); R21CA122270 (NIH)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — peginterferon alfa-2b; Decitabine

ARMS (2):
- Group 1 (chemotherapy) (Active Comparator): Patients receive decitabine IV over 1 hour on days 1-5 and 8-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients whose disease is not responding after the first course may crossover to group 2.
  Interventions: Drug: decitabine; Other: laboratory biomarker analysis
- Group 2 (chemotherapy and antineoplastic agent) (Experimental): Patients receive decitabine as in group 1 and pegylated interferon alfa-2b subcutaneously on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: peginterferon alfa-2b; Drug: decitabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: peginterferon alfa-2b — Given SC
  Other Names: PEG-IFN alfa-2b; pegylated interferon alfa-2b; polyethylene glycol IFN-A2b
  Arms: Group 2 (chemotherapy and antineoplastic agent)
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects of decitabine when given together with or without interferon alfa-2b, and the best dose of interferon alfa-2b, in treating patients with unresectable or metastatic solid tumors. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as interferon alfa-2b, may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether decitabine is more effective when given with or without interferon alfa-2b in treating solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess toxicities of decitabine plus escalating doses of pegylated interferon alfa-2b (PEG-Intron) in patients with metastatic solid tumor.

II. To identify the dose-limiting toxicity of decitabine in combination with escalating doses of pegylated interferon alfa-2b in these patients.

III. To identify the maximum tolerated dose of pegylated interferon alfa-2b in combination with decitabine in these patients.

SECONDARY OBJECTIVES:

I. To evaluate pretreatment and post-treatment blood and tumor samples to identify changes in global (genomic) DNA methylation.

II. To evaluate pretreatment and post-treatment blood, skin and tumor samples to identify changes in Mage-1 mRNA and protein expression, DNMT-1 levels (due to sequestration by 5-azacytidine), p53 induction (evidence of DNA damage response), as well as changes in levels of 2'5'-oligoadenylate synthesis, MxA and HLA class I as indicators of interferon response.

III. To evaluate complete and partial response rates in patients receiving decitabine in combination with escalating doses of pegylated interferon alfa-2b.

OUTLINE:

This is a dose-escalation study of pegylated interferon alfa-2b. Patients are assigned to 1 of 2 treatment groups.

GROUP 1 (control): Patients receive decitabine IV over 1 hour on days 1-5 and 8-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression after the first course of treatment may crossover to receive treatment in group 2.

GROUP 2: Patients receive decitabine as in group 1 and pegylated interferon alfa-2b subcutaneously on days 1, 8, 15, and 22.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample, normal skin, and tissue biopsy collection at baseline and periodically during study. Blood, normal skin, and tissue samples are analyzed for global (genomic) DNA methylation (gene-promoter methylation, gene and protein expression, p53 induction by DNA damage) and interferon levels by high-performance (pressure) liquid chromatography and PCR methylation assays, and for pharmacodynamic studies.

After completion of study treatment, patients are followed at 28 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven solid tumor

  * Metastatic or unresectable disease
* Tumor amenable to biopsy
* No curative or more effective treatment for this disease exists, in the opinion of the investigator
* Measurable disease by scans as assessed by RECIST criteria
* No untreated brain metastasis

  * No longer receiving steroid therapy for previously treated brain metastasis
* Zubrod performance status of 0-2
* Bilirubin ≤ 1.5 times upper limit normal (ULN)
* SGOT or SGPT ≤ 2.5 times ULN (≤ 5 ULN if hepatic metastases present)
* Serum creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* ANC > 1,500/μL
* Platelet count > 100,000/μL
* Hemoglobin > 9 g/dL (transfusion allowed)
* No NYHA class III-IV cardiac problems (e.g., congestive heart failure or myocardial infarction within the past 2 months)
* No severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, or active uncontrolled infection [e.g., HIV])
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study therapy
* Willing to undergo biopsies
* No medical or psychological conditions that, in the opinion of the investigator, may preclude the patient's ability to tolerate or complete the treatment, or to grant reliable informed consent
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I, II, or III cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* No prior extensive pelvic irradiation or prolonged nucleoside analogue pretreatment
* At least 28 days since prior and no concurrent chemotherapy, radiotherapy, surgery, biological therapy, anticancer agent, or other investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Toxicities as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 28 days
  The type, frequency, and severity of each toxicity will be reported.
Dose-limiting toxicity (DLT) of pegylated interferon alfa-2b when given with decitabine as assessed by NCI CTCAE version 3.0 | First 28-day course
  DLT is defined as grade III drug-related non hematologic and/or grade IV drug-related hematologic toxicity.
Maximum-tolerated dose (MTD) of pegylated interferon alfa-2b when given with decitabine as assessed by NCI CTCAE version 3.0 | First 28-day course
  The MTD will be the dose level where not more than 1 case of a specific grade III-IV drug-related toxicity is observed, and either 2+toxicities have been observed at the next highest dose level, or the maximum dose-level of PEG-Intron has been reached.

SECONDARY OUTCOMES:
Global (genomic) DNA methylation changes by high-performance liquid chromatography (HPLC) | Baseline to up to day 1 of course 2
  Repeated measures analysis of variance and other linear modeling techniques will be used.
Changes in expression of methylation-regulated genes in human biological tissues | Baseline to up to day 1 of course 2
  Repeated measures analysis of variance and other linear modeling techniques will be used.
Complete and partial response rates | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Samlowski, Principal Investigator — Nevada Cancer Institute-Summerlin Campus
Locations (1):
- Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada, United States